CLINICAL TRIAL: NCT02880358
Title: Epidemiology and Prognostic of the Acute Heart Failure in Northeast of France
Brief Title: Epidemiology and Prognostic of the Acute Heart Failure
Acronym: EPICAL2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 911069
Record Dates: First submitted 2013-07-31; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Decompensated Chronic Heart Failure; Heart Failure NYHA Class III; Acute Pulmonary Edema; Cardiogenic Shock; Heart Failure NYHA Class IV
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, whole blood and urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
EPICAL 2 (Epidemiology and prognostic of the Acute Heart Failure) is an epidemiological, observational, prospective and multicenter study. This study includes at first an exhaustive recording of the cases on a geographic area at East of France, then the recorded patients are followed up in a cohort at least 3 years. This study follows the experiences of the EPICAL study led by our team.

Main objective: To describe the characteristics of the patients affected by acute heart failure and to identify prognostic factors, in particular related to care. More exactly :

* To describe the sociodemographic, clinical, biological and therapeutic characteristics of the patients presenting an acute heart failure during hospitalisation and living at East of France ;
* To study the short and medium-term morbi-mortality of these patients, and identify the main factors determining the prognosis for survival ;
* To evaluate the prognostic impact of the intra and extra-hospital care ;
* To identify the evolution of the care's practices of the decompensated heart failure since the EPICAL study (15 years) and their influence on the prognosis of the disease.

Secondary objective: to constitute a biological collection of serum, plasma and urine of patients' sample presenting an acute heart failure.

DETAILED DESCRIPTION:
Criteria of inclusion:

* Patients hospitalized for acute heart failure or developing an acute heart failure during the hospitalisation in the intensive care, cardiology or geriatrics departments of the hospitals of Northeast of France during one year
* Patients died in emergencies or during the transfer, with a diagnosis of acute heart failure.

Acute heart failure includes decompensation of chronic heart failure, advanced stage of the heart failure, acute oedema of the lung and cardiogenic shock. According to the data of registers, the incidence of the acute heart failure in approximately 2,5 cases per 1000 adults per year, the expected sample size amounts to 2500 eligible patients over 1 year.

Data collection: the doctors declare the Acute Heart Failure of their departments. The technicians of clinical research collect the data concerning the sociodemographic, clinical, biological and therapeutic characteristics of the inclusive patients on arrival at the hospital, during the hospitalisation and at the exit. The biological takings are made for the patients having given their consent before the exit of the hospitalization. The patients are followed up during 3 years.

ELIGIBILITY:
Inclusion Criteria :

* Patients hospitalized for acute heart failure or developing an acute heart failure during the hospitalisation in the intensive care, cardiology or geriatrics departments of the hospitals of Northeast of France during one year
* Patients died in emergencies or during the transfer, with a diagnosis of acute heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute heart failure or developing an acute heart failure during the hospitalisation. It is an exhaustive recruitment in a region of Northeast of France. So, there is no sampling
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Acute Heart Failure | Inclusion

SECONDARY OUTCOMES:
Morbi-mortality of patients presenting an acute heart failure | Inclusion, 6 month, 1, 2 and 3 years after acute heart failure

OTHER OUTCOMES:
Effectiveness of therapeutic strategies on survival | Inclusion, 6 months, 1, 2, and 3 years after acute heart failure
  Patient medical record data (treatment, support network, therapeutic education)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Thilly, PU-PH, Principal Investigator — ¹ INSERM, CIC-EC, CIE6, Nancy, F-54 000, France ² CHU Nancy, Epidémiologie et Evaluation Cliniques, Nancy, F-54 000, France ³ Université de Lorraine, CIC-EC, CIE 6, Nancy, F-54 000, France
Locations (1):
- University Hospital Center, Nancy, Lorraine, France

REFERENCES:
- [Derived] Al-Gobari M, Agrinier N, Soudant M, Burnand B, Thilly N. Effects of Statins to Reduce All-Cause Mortality in Heart Failure Patients: Findings from the EPICAL2 Cohort Study. Am J Cardiovasc Drugs. 2019 Oct;19(5):497-508. doi: 10.1007/s40256-019-00346-4. PMID 30972619